CLINICAL TRIAL: NCT01775618
Title: A Multi-center, Phase III, Non-controlled, Open-label Trial to Evaluate the Pharmacokinetics, Safety, and Efficacy of BAY94-9027 for Prophylaxis and Treatment of Bleeding in Previously Treated Children (Age <12 Years) With Severe Hemophilia A
Brief Title: Safety and Efficacy of BAY94-9027 in Previously Treated Male Children With Haemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15912; 2012-004434-42 (EudraCT Number)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Factor VIII; Prophylaxis; Pediatric
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Main study (Experimental): Participants were treated and prophylaxis administered with BAY94-9027 at a dose of 25-60 international units/kilogram (IU/kg) twice per week or 45-60 IU/kg every 5 days or 60 IU/kg every 7 days as an intravenous (IV) infusion as per clinical needs of each subject up to at least 50 exposure days (EDs) and a minimum of at least 6 months.
  Interventions: Biological: BAY94-9027
- Part 2 (Expansion group) (Experimental): Participants were administered with BAY94-9027 at a dose of 25-60 IU/kg twice per week for prophylaxis for 12 weeks.
  Interventions: Biological: BAY94-9027
- Extension study (Experimental): Participants were treated and prophylaxis administered with BAY94-9027 at a dose of 25- 60 IU/kg twice per week or 45-60 IU/kg every 5 days or 60 IU/kg every 7 days as an IV infusion as per clinical needs of each subject for at least 50 EDs or until marketing authorization of the drug.
  Interventions: Biological: BAY94-9027

INTERVENTIONS:
Biological: BAY94-9027 — Study drug dosing was adjusted to the clinical needs of each subject in the range of 25-60 IU/kg/administration, intravenous infusion, at least 50 EDs and a minimum of at least 6 months
  Arms: Main study
Biological: BAY94-9027 — Twice per week prophylaxis: 25-60 IU/kg, intravenous infusion, for 12 weeks
  Arms: Part 2 (Expansion group)
Biological: BAY94-9027 — Study drug dosing was adjusted to the clinical needs of each subject in the range of 25-60 IU/kg/administration, intravenous infusion, at least 50 additional EDs to achieve at least 100 cumulative EDs, or until marketing authorization of the drug
  Arms: Extension study

SUMMARY:
Hemophilia A is an inherited blood disorder in which one protein, Factor VIII, needed to form blood clots is missing or not present in sufficient levels. Hemophilia A causes the clotting process to be slowed and the person experiences bleeds causing serious problems that could lead to disability. The current standard treatment for severe hemophilia A is infusion of FVIII to stop bleeding, or regular scheduled treatment to prevent bleeds from occuring. Due to the short half-life of FVIII, prophylaxis may require treatment as often as every other day.

In this trial safety and efficacy of a long-acting recombinant Factor VIII molecule is being evaluated in 50 male subjects, < 12 years of age, with severe Hemophilia A. These subjects will receive open label treatment with long-acting rFVIII for approximately 6 months (or longer until 50 exposure days) on a regular schedule at least once every 7-days. Doses and dose intervals may be adapted to the subject's clinical need. A second group of patients will receive open label treatment with the same drug for 12 weeks on a regular schedule of 2x/week. Patients will attend the treatment center for routine blood samples and will be required to keep an electronic diary.

Subjects will be offered participation in an optional extension study to collect observations for at least an additional 50 exposure days.

ELIGIBILITY:
Inclusion Criteria:

* Males < 12 years of age
* Subjects with severe hemophilia A
* Previously treated with FVIII for > 50 exposure days

Exclusion Criteria:

* Subjects with current evidence of or history of inhibitors to FVIII
* Any other inherited or acquired bleeding disorder
* Platelet counts < 100,000/mm^3
* Creatinine > 2x the upper limit of normal
* Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) > 5x the upper limit of normal

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Annualized number of all bleeds | At least 50 exposure days (ED) over 6 months, on average 245 days
Pharmacokinetics profile of BAY94-9027 based on blood concentration over the defined time period | Pre-dose to 72 hours post-dose
  Pharmacokinetics profile includes maximum concentration (Cmax), half-life (t1/2), area under the concentration versus time curve (AUC), mean residence time (MRT), volume of distribution at steady state (Vss), and clearance (CL)
Response of acute bleeding events to treatment based on a 4-point scale (poor, moderate, good, or excellent) | At least 50 exposure days (ED) over 6 months, on average 245 days
Characterization of a potential immune response | 12 weeks
Inhibitor development in the extension study | At least 50 additional EDs to achieve at least 100 cumulative EDs, on average 5 years

SECONDARY OUTCOMES:
Inhibitor development in the main study | After 10 to 15 and 50 exposure days (ED) over 6 months, on average 245 days
Assessment of incremental recovery in main study | At least 50 exposure days (ED) over 6 months, on average 245 days
Number of participants with adverse events as a measure of safety and tolerability | From the start of study treatment up to 7 days after the last dose (Main study: on average 245+7 days; Part 2: 12 weeks+7 days; Extension study: on average 5 years+7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- United States (7):
  - Sacramento, California
  - Pensacola, Florida
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Salt Lake City, Utah
- La Plata, Buenos Aires, Argentina
- Vienna, Austria
- Belgium (2):
  - Ghent
  - Leuven
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Canada (2):
  - Calgary, Alberta
  - Toronto, Ontario
- Thessaloniki, Greece
- Ramat Gan, Israel
- Italy (3):
  - Milan, Lombardy
  - Palermo, Sicily
  - Padua, Veneto
- Vilnius, Lithuania
- Netherlands (2):
  - Amsterdam
  - Utrecht
- New Zealand (2):
  - Christchurch
  - Hamilton
- Oslo, Norway
- Poland (2):
  - Lodz
  - Olsztyn
- Romania (2):
  - Bucharest
  - Timișoara
- Esplugues de Llobregat, Barcelona, Spain
- United Kingdom (4):
  - Newcastle upon Tyne, Tyne and Wear
  - Bristol
  - Manchester
  - Sheffield

REFERENCES:
- [Derived] Mancuso ME, Biss T, Fischer K, Maas Enriquez M, Steele M, Wang M, Tseneklidou-Stoeter D, Ahuja S, Kenet G. PROTECT VIII kids extension study: Long-term safety and efficacy of BAY 94-9027 (damoctocog alfa pegol) in children with severe haemophilia A. Haemophilia. 2021 May;27(3):434-444. doi: 10.1111/hae.14294. Epub 2021 Mar 16. PMID 33724632
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — https://www.clinicaltrialsregister.eu/